CLINICAL TRIAL: NCT05013879
Title: Effect of Kinesiotaping on Edema Management, Pain and Function on Patients With Bilateral Total Knee Arthroplasty
Brief Title: Kinesiotape for Edema After Bilateral Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Burke Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13203
Record Dates: First submitted 2021-08-02; First posted 2021-08-19 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty Complications; Arthroplasty, Replacement, Knee
Keywords: edema; arthroplasty, knee, bilateral; kinesiotaping
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: Repeated measures with two within-subjects factors: time and taped/untaped leg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape leg plus standard rehabilitation (Experimental): Kinesio(R)Tape for edema management applied to a randomly selected lower extremity plus standard inpatient rehabilitation after bilateral total knee arthroplasty
  Interventions: Device: Kinesio(R)Tape for edema control
- Control leg with standard rehabilitation alone (No Intervention): Control leg receiving standard inpatient rehabilitation alone.

INTERVENTIONS:
Device: Kinesio(R)Tape for edema control — Kinesio(R)Tape is an elastic, cotton tape with an adhesive backing. When applied for edema management, strips of Kinesio(R)Tape are applied to the lower leg in a criss-cross fashion by a physical therapist who is a Certified Kinesiotape Practitioner.
  Other Names: kinesiotaping or kinesiological taping
  Arms: Kinesiotape leg plus standard rehabilitation

SUMMARY:
The purpose of this study is to determine if kinesiotaping for edema management will decrease post-operative edema in patients with bilateral total knee arthroplasty. The leg receiving kinesiotaping during inpatient rehabilitation may have decreased edema and pain and improved movement and function when compared to the leg not receiving kinesiotape.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients undergoing inpatient rehabilitation after bilateral total knee arthroplasty will have Kinesio(R)Tape applied to one randomly selected leg while the other leg serves as a control. Measurement of bilateral leg circumference, knee range of motion, numerical rating scale for pain, and selected questions from the Knee Injury and Osteoarthritis Outcome Score will occur at regular intervals throughout the rehabilitation stay. Patients will receive standard rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* admitted to Burke Rehabilitation Hospital for inpatient rehabilitation within 5 days after same-day or staged bilateral total knee arthroplasty;
* 50-85 years of age;
* able to read and understand English or a hospital-provided translator when consenting for the study;
* free from contraindications for kinesiotaping (see below); and,
* able to tolerate an active rehabilitation program.

Exclusion Criteria:

* stage III or IV heart failure, stage III or IV renal failure;
* fragile, very hairy or sensitive skin;
* anesthesia or paraesthesia of any area of the lower extremity, except the surgical sites
* active skin rashes or infections or skin lesions in the lower extremity;
* prior history of allergic reactions to skin taping, bandaids, surgical tape; athletic tape or other skin-adhering electrode adhesives;
* prior history of lower extremity lymphedema;3
* prior history of lower extremity venous or arterial disease;
* post-operative complications in the surgical sites;4
* partial joint arthroplasty or revision arthroplasty of one or both knees;1,5
* inability to give informed consent offered in English or through a hospital-provided translator
* age less than 50 years or over 85 years;
* inability to tolerate an active rehabilitation program.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline and during 1-2-day time intervals of circumferences of both knees and lower extremities | During inpatient rehabilitation stay for each subject: at baseline (day 0), day 1, day 2, and every other day until day 8
  Bilateral circumferences, in centimeters, at the following points: 10 cm above the superior pole of the patella; middle of the knee joint; calf circumference at the broadest part of the calf and at 3 inches below the fibular head landmark; figure of eight method for foot and ankle circumference - a measurement from the lateral malleolus to the navicular tuberosity, under the plantar aspect of the foot towards the tuberosity of the fifth metatarsal, around to the medial malleolus, and posterior to the leg to return to the lateral malleolus.

SECONDARY OUTCOMES:
Change from baseline and day-to-day changes of bilateral knee pain on numerical pain rating scale | During inpatient rehabilitation stay for each subject: at baseline (day 0), day 1, day 2, and every other day until day 8
  Patient self-report: Pain rating for each leg on a integer scale of 0 (no pain) to 10 (worst pain imaginable)
Change from baseline and during 1-2-day time intervals for bilateral knee range of motion | During inpatient rehabilitation stay for each subject: at baseline (day 0), day 1, day 2, and every other day until day 8
  Physical therapist's measurement of active and active assistive knee range of motion (degrees) for flexion and extension using a standard goniometer
Change from baseline to Day 4 to Discharge Day for selected parts of the Knee Injury and Osteoarthritis Outcome Score (KOOS) self-report | At start of study, 4 days after start of study, and day 8
  Patient self-report using the KOOS sections relating to pain, stiffness, activities of daily living
Change from baseline and during 1-2-day time intervals for Timed Up-and-Go Test | During inpatient rehabilitation stay for each subject: at baseline (day 0), day 1, day 2, and every other day until day 8
  Time (sec) to rise from a seated position, walk 10 m, turn, walk back to seat, and sit down. Patient will use appropriate assistive device and have appropriate guarding by a physical therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Babyar, PT, PhD, Principal Investigator — Burke Rehabilitation Hospital
Locations (1):
- Burke Rehabilitation Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tornatore L, De Luca ML, Ciccarello M, Benedetti MG. Effects of combining manual lymphatic drainage and Kinesiotaping on pain, edema, and range of motion in patients with total knee replacement: a randomized clinical trial. Int J Rehabil Res. 2020 Sep;43(3):240-246. doi: 10.1097/MRR.0000000000000417. PMID 32459670
- [Background] Guney Deniz H, Kinikli GI, Onal S, Sevinc C, Caglar O, Yuksei I. Comparison of Kinesio Tape application and manual lymphatic drainage on lower extremity oedema and functions after total knee arthroplasty. [Abstract]. Ann Rheum Dis. 2018; 77: 1791.
- [Background] Donec V, Krisciunas A. The effectiveness of Kinesio Taping(R) after total knee replacement in early postoperative rehabilitation period. A randomized controlled trial. Eur J Phys Rehabil Med. 2014 Aug;50(4):363-71. Epub 2014 May 13. PMID 24819349
- [Background] Sulman M, Riaz S, Khan RR, Faisal Z, Rajput R, Noor M. Effectiveness of Kinesio Taping on pain and function after total knee arthroplasty. Pak J Med Health Sci. 2020;14:1267-1270.
- [Background] Oktas B, Vergili O. The effect of intensive exercise program and kinesiotaping following total knee arthroplasty on functional recovery of patients. J Orthop Surg Res. 2018 Sep 12;13(1):233. doi: 10.1186/s13018-018-0924-9. PMID 30208939
- [Background] Alghadir A, Anwer S, Brismee JM. The reliability and minimal detectable change of Timed Up and Go test in individuals with grade 1-3 knee osteoarthritis. BMC Musculoskelet Disord. 2015 Jul 30;16:174. doi: 10.1186/s12891-015-0637-8. PMID 26223312
- [Background] Hancock GE, Hepworth T, Wembridge K. Accuracy and reliability of knee goniometry methods. J Exp Orthop. 2018 Oct 19;5(1):46. doi: 10.1186/s40634-018-0161-5. PMID 30341552
- [Background] Unver B, Ertekin O, Karatosun V. Pain, fear of falling and stair climbing ability in patients with knee osteoarthritis before and after knee replacement: 6 month follow-up study. J Back Musculoskelet Rehabil. 2014;27(1):77-84. doi: 10.3233/BMR-130422. PMID 23948839
- [Background] Bakar Y, Ozdemir OC, Sevim S, Duygu E, Tugral A, Surmeli M. Intra-observer and inter-observer reliability of leg circumference measurement among six observers: a single blinded randomized trial. J Med Life. 2017 Jul-Sep;10(3):176-181. PMID 29075347
- [Background] Collins NJ, Roos EM. Patient-reported outcomes for total hip and knee arthroplasty: commonly used instruments and attributes of a "good" measure. Clin Geriatr Med. 2012 Aug;28(3):367-94. doi: 10.1016/j.cger.2012.05.007. Epub 2012 Jun 22. PMID 22840304
- [Derived] DalCeredo C, LaCava J, Young R, Conklin K, Herbold J, Simsuangco C, Inostroza Millas F, Sokolow Z, Babyar S. Effectiveness of kinesiotaping for lymphatic drainage after bilateral total knee arthroplasty: A randomized controlled trial. Medicine (Baltimore). 2025 Apr 11;104(15):e41971. doi: 10.1097/MD.0000000000041971. PMID 40228285